CLINICAL TRIAL: NCT02033603
Title: A Randomised Controlled Trial Comparing Single Shot Adductor Canal Block With Femoral Nerve Block for Analgesia Post Total Knee Arthroplasty
Brief Title: Adductor Canal Versus Femoral Nerve Block for Analgesia Post Total Knee Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/ 921/ D
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-01

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty; Total knee replacement; Femoral Nerve Block; Adductor Canal Block
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral Nerve Block (Active Comparator): Femoral Nerve block performed with 0.5% Ropivacaine 30mls (150mg)
  Interventions: Drug: Ropivacaine
- Adductor Canal block (Active Comparator): Adductor Canal block performed with 0.5% Ropivacaine 30mls (150mg)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — 30mls of 0.5% ropivacaine
  Other Names: naropin

SUMMARY:
Total knee arthroplasty or replacement (TKA) is a surgery performed for osteoarthritis of the knee which is increasingly performed as the population ages. It is a painful surgery and one of the methods to reduce post-operative pain is performing a regional anaesthesia technique. The current practice is to perform a femoral nerve block (FNB) which blocks the nerves supplying the knee joint and the thigh muscles (quadriceps). This provides effective analgesia. However, it also results in weakness of the quadriceps and may result in falls post-operatively.

Adductor canal block (ACB) is a new, alternative regional anaesthesia technique which is hypothesised to provide as effective analgesia, with less quadriceps weakness compared to FNB, hence potentially reducing the risk of falls post-operatively.

Investigators aim to study if the analgesia provided by ACB is as good as FNB while preserving quadriceps strength.

ELIGIBILITY:
Inclusion Criteria:

* ages 45-85
* American Society of Anaesthesiologists physical status 1-3
* BMI 18-35 kg/m2

Exclusion Criteria:

* inability to give consent, communicate, cooperate
* Patients with regular consumption of strong opioids (morphine, oxycodone) or steroids
* Patients with allergy to local anaesthetics or any drugs included in the study
* Patients with lower limb surgery in the preceding year
* Patients with pre-existing neurological deficits
* Patients who are unsuitable for general anaesthetics (eg difficult airway)

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | first 24 hours

SECONDARY OUTCOMES:
Pain scores | 1, 6, 12, 24, 48
Morphine consumption | 48 hours
Side effects of opioids- sedation, nausea and vomiting | 48 hours
Quadriceps strength, ability to mobilise | 24, 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yean Chin Lim, MBBS, MMed, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore